CLINICAL TRIAL: NCT00541307
Title: Post Marketing Study of the GORE VIABAHN Endoprosthesis With Heparin Bioactive Surface in the Treatment of Superficial Femoral Artery Obstructive Disease (VIPER)
Brief Title: GORE VIABAHN Endoprosthesis With Heparin Bioactive Surface in the Treatment of SFA Obstructive Disease (VIPER)
Acronym: VIPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VPR 07-03
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-11

CONDITIONS: Peripheral Vascular Diseases
Keywords: Peripheral Arterial Disease; Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GORE VIABHAN Endoprothesis (Experimental): Treatment with the GORE VIABAHN Endoprosthesis with Heparin Bioactive Surface
  Interventions: Device: Treatment with the GORE VIABAHN Endoprosthesis with Heparin Bioactive Surface

INTERVENTIONS:
Device: Treatment with the GORE VIABAHN Endoprosthesis with Heparin Bioactive Surface — Endovascular treatment of the study lesion with the GORE VIABAHN Endoprosthesis with Heparin Bioactive Surface

SUMMARY:
The objective of the study is collect data on the GORE VIABAHN Endoprosthesis with Heparin Bioactive Surface in the treatment of chronic Superficial Femoral Artery disease. Device patency at 12 months is the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:>

* lifestyle limiting claudication, rest pain or minor tissue loss>
* ABI (ankle-brachial index) < 0.9 or TBI (toe-brachial index) < 0.5 if ABI is >0.9
* Stenosis (>50%) or occlusion of native SFA (superficial femoral artery) >5cm
* Orifice and 1 cm of SFA are patent
* Popliteal artery is patent at the intercondylar fossa of the femur to the trifurcation
* At least 1 patent run off vessel
* Guidewire and deliver system successfully traversed the lesion

Exclusion Criteria:>

* Untreated flow-limiting aortoiliac occlusive disease
* Any previous stenting or surgery in the target vessel
* Femoral or popliteal aneurysm of target vessel
* No patent tibial arteries
* Prior ipsilateral femoral artery bypass
* Major distal amputation (above the transmetatarsal) in either limb
* Patients with known sensitivity to Heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Saxon, MD, Principal Investigator — North County Radiology Medial Group Inc.
Locations (5):
- United States (5):
  - Tri-City Medical Center, Oceanside, California
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Columbia Surgical Associates, Columbia, Missouri
  - Baylor University Medical Center, Dallas, Texas
  - St. Luke's Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Gore Viabahn Endoprosthesis: All patients enrolled in this single arm study were treated with the Gore Viabahn Endoprosthesis.
Period: Overall Study
Arm/Group | Gore Viabahn Endoprosthesis
Started | 119
Completed | 95
Not Completed | 24
Not completed — Death | 5
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 4
Not completed — Subject returned early (outside window) | 1
Not completed — Surgical Bypass | 5

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Subjects: The total number of enrolled subjects.
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 61
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 74
Region of Enrollment [Number; unit: participants]
  United States | 119

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency at 12 Months
Description: Primary patency is defined as no evidence of restenosis (repeat narrowing) or occlusion (total blockage) within the originally treated lesion based on color-coded duplex sonography (color Doppler ultrasound (CDUS). The Peak Systolic Velocity Ratio must be less than 2.5 (PSVR: the result of taking the highest rate of blood flow within the stented region and dividing it by the highest rate of blood flow just above the stented area).
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Gore Viabahn Endoprosthesis
Number analyzed (Participants) | 119
percentage of subjects | 72.9 [62.9 to 80.6]

2. Secondary Outcome: Proportion of Subjects Who Experience Major Device-related Adverse Events Within the First 30 Days
Description: If the functioning or characteristics of the device caused or contributed significantly to the adverse event,and if they occurred within 30 days of the procedure, they would be considered major adverse events (MAEs). Major AEs require significant therapy, including an unplanned increase in the level of care, permanent sequelae, hospitalization, or death.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Gore Viabahn Endoprosthesis
Number analyzed (Participants) | 119
participants | 0

3. Secondary Outcome: Primary Assisted Patency
Description: Primary assisted patency is defined as patency in the target lesion maintained by repeat intervention (one or more follow-up procedures) in an attempt to salvage the stent prior to complete occlusion (blockage) of the treated arterial segment, and also includes patients with primary patency.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Gore Viabahn Endoprosthesis
Number analyzed (Participants) | 119
percentage of subjects | 85.6 [77.2 to 91.1]

4. Secondary Outcome: Secondary Patency
Description: Secondary patency is defined as patency in the target lesion maintained by repeat intervention (one more more follow-up procedures) after complete occlusion (blockage) of the treated arterial segment, and also includes patients that have primary and primary assisted patency.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Gore Viabahn Endoprosthesis
Number analyzed (Participants) | 119
percentage of subjects | 92.2 [84.9 to 96.0]

5. Secondary Outcome: Device-related Major Adverse Events at 12 Months
Description: If the functioning or characteristics of the device caused or contributed significantly to the adverse event (AE), the AE would be related to the device. Major AEs require significant therapy, including an unplanned increase in the level of care, permanent sequelae, hospitalization, or death.
Time Frame: 12 months
Measure: Number; unit: event
Arm/Group | Gore Viabahn Endoprosthesis
Number analyzed (Participants) | 119
event | 1

ADVERSE EVENTS:
Groups:
- Gore VIABAHN Endoprosthesis With Heparin Bioactive Surface: Gore VIABAHN Endoprosthesis with Heparin Bioactive Surface
Arm/Group | Gore VIABAHN Endoprosthesis With Heparin Bioactive Surface
Serious Adverse Events (participants affected / at risk) | 11/119
Other Adverse Events (participants affected / at risk) | 0/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gore VIABAHN Endoprosthesis With Heparin Bioactive Surface (N=119)
Acute myocardial infarction, unspecified site (Cardiac disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Chronic renal failure (Renal and urinary disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Claudication (Vascular disorders) | 1 (1)
Femoral artery embolism (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Ischemic leg ulcer (Vascular disorders) | 1 (1)
Thrombosis in device (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator will provide the materials to the sponsor at least 30 days in advance of submission for publication or public disclosure. The sponsor has the right to make modifications as necessary to protect proprietary information or correct inaccuracies in technical specifications or device descriptions.